CLINICAL TRIAL: NCT01707381
Title: A Randomized, Single-Center, Open-Label, Crossover Study Comparing the Efficacy of BOL-303259-X Ophthalmic Solution With Timolol Maleate Ophthalmic Solution 0.5% in Subjects With Open-Angle Glaucoma or Ocular Hypertension.
Brief Title: BOL-303259-X With Timolol 0.5% in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Acronym: Constellation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 803
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Ocular Hypertension; Open Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — BOL 303259-X; Timolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Timolol Maleate (Active Comparator): Timolol maleate ophthalmic solution 0.5% administered 1 drop BID once in morning and once in the evening for 4 weeks.
  Interventions: Drug: Timolol maleate
- BOL-303259-X (Experimental): BOL-303259-X topical ophthalmic solution administered 1 drop QD in the evening for 4 weeks.
  Interventions: Drug: BOL-303259-X

INTERVENTIONS:
Drug: BOL-303259-X — Topical ophthalmic solution
  Arms: BOL-303259-X
Drug: Timolol maleate — Topical ophthalmic solution
  Arms: Timolol Maleate

SUMMARY:
This clinical investigation is being performed to compare the effect of BOL-303259-X dosed once daily (QD) with timolol maleate 0.5% dosed twice daily (BID) in reducing intraocular pressure (IOP) measured over a 24-hour period in subjects with open-angle glaucoma (OAG) or ocular hypertension (OHT).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of OAG or OHT in 1 or both eyes.
* Subjects who are treatment-naïve must meet the following IOP requirements at Visit 1 (Screening), and pretreated subjects must meet the following IOP requirements at Visit 2 (Washout): Intraocular pressure ≥ 22 mmHg in at least 1 eye and ≤ 36 mmHg in both eyes.

Exclusion Criteria:

* Subjects who have been exposed to BOL-303259-X within 3 months prior to Visit 1 (Screening).
* Subjects with a history or presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the subject or confound the results of the study.
* Subjects with an irregular daily sleep schedule.
* Subjects who are unable to wear sleep monitoring device for 7 days prior to laboratory study.
* Subjects with an anticipated need to initiate or modify medication (systemic or topical) that is known to affect IOP.
* Subjects for whom concomitant use of medications may interact with the safety or efficacy of a nitric oxide.
* Subjects with known hypersensitivity or contraindications to latanoprost or any of the ingredients in the study drugs.
* Subjects who are expected to require treatment with ocular or systemic corticosteroids.
* Subjects who are in need of any other topical or systemic treatment of OAG or OHT.
* Subjects who are unable to discontinue contact lens use during and for 24 hours before the laboratory study.
* Subjects with a central corneal thickness greater than 600 μm in either eye.
* Subjects with any condition that prevents reliable applanationtonometry in either eye.
* Subjects with advanced glaucoma and subjects with a cup/disc ratio greater than 0.8 or a history of split fixation, or a field loss threatening fixation in either eye.
* Subjects with previous or active corneal disease.
* Subjects with a history of severe dry eye.
* Subjects with active optic disc hemorrhage.
* Subjects with a history of central/branch retinal vein or artery occlusion.
* Subjects with a history of macular edema.
* Subjects with very narrow angles and subjects with angle closure, congenital, and secondary glaucoma, and subjects with history of angle closure in either eye.
* Subjects with a diagnosis of a clinically significant or progressive retinal disease in either eye.
* Subjects with any intraocular infection or inflammation within 3 months prior to Visit 1 (Screening).
* Subjects with a history of ocular laser surgery within the 3 months prior to Visit 1 (Screening).
* Subjects with a history of incisional ocular surgery or severe trauma within 3 months prior to Visit 1 (Screening).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quintus Ngumah, OD, PhD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- University of California San Diego, La Jolla, California, United States

REFERENCES:
- [Result] Liu JHK, Slight JR, Vittitow JL, Scassellati Sforzolini B, Weinreb RN. Efficacy of Latanoprostene Bunod 0.024% Compared With Timolol 0.5% in Lowering Intraocular Pressure Over 24 Hours. Am J Ophthalmol. 2016 Sep;169:249-257. doi: 10.1016/j.ajo.2016.04.019. Epub 2016 Jul 22. PMID 27457257

RESULTS

PARTICIPANT FLOW:
Groups:
- Timolol Maleate Cross Over to BOL-303259X: Participants first recieved timolol maleate ophthalmic solution 0.5% administered 1 drop BID once in morning and once in the evening for 4 weeks. Thereafter they received BOL-303259X once in the evening for 4 weeks.
- BOL-303259-X Crossover to Timolol Maleate: Participants first received BOL-303259-X topical ophthalmic solution administered 1 drop QD in the evening for 4 weeks. Thereafter, they received timolol maleate ophthalmic solution 0.5% administered 1 drop BID once in morning and once in the evening for 4 weeks.
Period: Period 1
Arm/Group | Timolol Maleate Cross Over to BOL-303259X | BOL-303259-X Crossover to Timolol Maleate
Started | 12 | 13
Completed | 10 | 11
Not Completed | 2 | 2
Period: Period 2
Arm/Group | Timolol Maleate Cross Over to BOL-303259X | BOL-303259-X Crossover to Timolol Maleate
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population: All randomized subjects who received at least one dose of study drug, had a baseline and at least one postbaseline intraocular assessment.
Groups:
- All Study Participants: Participants who were randomized to receive either latanoprostene ophthalmic solution 0.024% or timolol maleate 0.5%
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Treatment-Naive [Count of Participants; unit: Participants] | 15

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour IOP
Description: Supine intraocular pressure (IOP) measured in the study eye following 4 weeks of treatment
Time Frame: after 4 weeks of treatment
Population: Intent to Treat (ITT) Population:All randomized subjects who received at least one dose of study drug, had a baseline and at least one postbaseline intraocular assessment.
Measure: Least Squares Mean (Standard Deviation); unit: mm Hg
Arm/Group | Timolol Maleate | BOL-303259-X
Number analyzed (Participants) | 21 | 21
mm Hg | 23.55 (2.46) | 21.77 (2.37)
Statistical Analysis 1: Comparison: Timolol Maleate vs BOL-303259-X; Test type: Other; p < 0.001, ANCOVA; Treatment difference = -1.773, 95% CI 2-sided [-2.380 to -1.166] — Treatment Difference = BOL-303259-X 0.024% - Timolol maleate 0.5%

2. Secondary Outcome: 24-hour Ocular Perfusion Pressure
Description: Sitting Ocular Perfusion Pressure = 95/140 x mean arterial blood pressure - IOP; Supine Ocular Perfusion Pressure = 115/130 x mean arterial blood pressure - IOP; the nocturnal time frame encompassed measures taken at 10pm, 12am, 2am and 4 am; whereas the diurnal time frame encompassed measures taken at 6am, 8am, 10am, 12pm, 2pm, 4pm, 6pm, and 8pm.
Time Frame: after 4 weeks of treatment
Population: Intent to Treat (ITT): All randomized subjects who received at least one dose of study drug, had a baseline, and at least one post baseline intraocular assessment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Timolol Maleate | BOL-303259-X
Number analyzed (Participants) | 21 | 21
mm Hg
  OPP (nocturnal) | 48.4 (9.4) | 52.5 (9.5)
  OPP (Diurnal supine) | 54.8 (7.5) | 55.9 (7.8)
  OPP (Diurnal sitting) | 43.2 (5.7) | 45.2 (6.8)
Statistical Analysis 1: Comparison: Timolol Maleate vs BOL-303259-X; Statistical analysis of nocturnal (supine) OPP was performed among baseline, the BOL-303259-X treatment and timolol treatment using ANOVA. the criteria for statistical significance was P<0.05. Post hoc Bonferroni T-tests were then utilized to compare BOL and timolol groups; Test type: Other; p < 0.05, ANOVA; Bonferroni t-test used for paired compar = 0.010 — the bonferroni result applies to nocturnal supine OPP data comparing BOL group to timolol group

3. Secondary Outcome: IOP Area Under the Curve Over 24 Hours
Description: The Area Under the Curve(AUC) is the weighted average of IOP over all 24-hour IOP assessment times (2pm, 4pm, 6pm, 8pm, 10pm, 12am, 2am, 4am, 6am, 8am, 10am, 12pm). The AUC was calculated using the trapezoidal rule.
Time Frame: after 4 weeks of treatment
Population: ITT population
Measure: Least Squares Mean (Standard Deviation); unit: mm Hg
Arm/Group | Timolol Maleate | BOL-303259-X
Number analyzed (Participants) | 21 | 21
mm Hg | 23.54 (2.44) | 21.77 (2.29)
Statistical Analysis 1: Comparison: Timolol Maleate vs BOL-303259-X; Test type: Other; p = 0.004, ANOVA; Mean Difference (Final Values) = -1.770, 95% CI 2-sided [-2.915 to -0.625] — Treatment Difference = BOL-303259-X 0.024% - Timolol maleate 0.5%

ADVERSE EVENTS:
Time Frame: Four weeks for each intervention
Description: Safety population included all participants who received at least one dose of intervention
Arm/Group | Timolol Maleate | BOL-303259-X
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 4/23 | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Timolol Maleate (N=23) | BOL-303259-X (N=23)
Punctate keratitis (Eye disorders) | 3 | 0
Instillation site erythema (General disorders) | 0 | 1
Instillation site irritations (General disorders) | 1 | 0
Dizziness (Cardiac disorders) | 1 | 0
Dyspnoea (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
hyperhidrosis (General disorders) | 0 | 1
Blood pressure decreased (Investigations) | 1 | 0
Heart rate decreased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No